CLINICAL TRIAL: NCT03929120
Title: A Phase I Study to Evaluate the Safety of Allogeneic Bone Marrow Derived Mesenchymal Stem Cells for Interstitial Lung Disease in Patients With Connective Tissue Disorders
Brief Title: Allogeneic Bone Marrow Mesenchymal Stem Cells for Patients With Interstitial Lung Disease (ILD) & Connective Tissue Disorders (CTD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Andy Abril, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-007216
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Interstitial Lung Disease; Connective Tissue Diseases
MeSH Terms: conditions — Lung Diseases, Interstitial; Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Interstitial Lung Disease with Connective Tissue Disorder (Experimental): Subjects with Interstitial Lung Disease (ILD) associated with Connective Tissue Disorder (CTD) will receive a new treatment called Allogeneic (coming from a healthy donor) Bone Marrow Derived Mesenchymal Stem Cells (BMD-MSCs)
  Interventions: Biological: Allogeneic Bone Marrow Derived Mesenchymal Stem Cells (BMD-MSCs)

INTERVENTIONS:
Biological: Allogeneic Bone Marrow Derived Mesenchymal Stem Cells (BMD-MSCs) — Subjects will be treated with regular standard of care plus 0.5-1 million MSC/Kg intravenously.

SUMMARY:
Researchers are trying to find out more about the safety of a new treatment, Allogeneic (coming from a healthy donor) Bone Marrow Derived Mesenchymal Stem Cells (BMD-MSCs) which is still experimental, for Interstitial Lung Disease (ILD) associated with Connective Tissue Disorder (CTD).

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age and less than 80 years of age
* Both female and male
* Patients with new diagnosis of interstitial lung disease associated with connective tissue disorders, Antineutrophil cytoplasmic antibodies (ANCA) associated vasculitis or idiopathic pneumonia with autoimmune features (IPAF) or established diagnosis of ILD associated with CTD under conventional therapy for at least 6 months but less than 24 months, with no evidence of improvement.
* Competent and able to provide written informed consent, and ability to comply with protocol

Exclusion Criteria:

* Patients with interstitial lung disease without evidence of a concomitant rheumatologic autoimmune disorder
* Exposure to rituximab or cyclophosphamide on the previous 2 months
* Severe interstitial lung disease defined by the presence of severe hypoxemia at rest (SO2 < 88% at rest)
* Clinical assessment that indicates active chronic infections such as osteomyelitis or active tuberculosis (TB), or acute infections such as pneumonia, active bronchitis, cellulitis, etc. or active solid tumors or hematologic malignancies
* Previous treatment with mesenchymal stem cells
* Clinically significant medical conditions within the six months before administration of BMD-MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
* Medical history of human immunodeficiency virus (HIV), Hepatitis B or C
* Abnormal complete blood count (CBC), creatinine, Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) at screening
* Pregnant or breast feeding
* Unwilling to agree to use acceptable contraception methods during participation in the trial
* Inability to provide informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 6 months
  Number of adverse events reported with infusion of each intravenous Mesenchymal Stem Cells (MSC) dose

CONTACTS AND LOCATIONS:
Overall Officials: Andy Abril, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials